CLINICAL TRIAL: NCT01997697
Title: Predictive Factors of the Reduction of Emotional Eating After a Behavior Change Program Among Individuals With Obesity of Class II and Class III.
Brief Title: Reduction of Emotional Eating After a Behavior Change Program in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9110
Record Dates: First submitted 2013-11-21; First posted 2013-11-28 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with obesity (Experimental): behavior change program among patients with obesity
  Interventions: Other: behavior change program

INTERVENTIONS:
Other: behavior change program — behavior change program among patients with obesity

SUMMARY:
Recent studies show that overweight people have a greater sensitivity to the rewarding aspect of food due to the disturbance of the dopaminergic system. These perturbations lead to a greater amount of food to satisfy this rewarding aspect. Then, this rewarding aspect to food would also facilitate food intake related to emotions, whether they are positive or negative. However, the food intake in response to emotions can be modulated by physical activity. But, there are no interventional studies in the literature examining the behavioral and biological factors related to emotional eating together with the fact, there are few data on the explanatory mechanisms. The purpose of the study is to evaluate the predictive factors of emotional eating 6 months after a behavior change program adapted to the motivational state and to identify the its underlying mechanisms

DETAILED DESCRIPTION:
While emotional eating, food intake in response to emotions, can be modulated by physical activity, the practice of that latter is difficult mostly in people with overweight. Thus, there is a need to adapt the practice of physical activity in function of the motivation of the individual. One of most prominent theoretical model is the transtheoretical model. Regarding changes in physical activity and eating behavior, some data suggest that the processes of change from the transtheoretical model predict the efficacy of a treatment and thus its therapeutic success. The motivational approach could lead to self-regulation of emotions and therefore a decrease in emotional eating. Methods The study is a prospective cohort. Participants are exposed to a five-days hospitalization and engaged in a program of therapeutic education. During this hospitalization, there are some collective and individuals workshop on topics related to physical activity and nutrition. Intervention The intervention is based on the processes of change from the transtheoretical model. There are 5 experiential and 5 behavioral processes of change. Thus, according to the response of a questionnaire evaluating these processes of change, participants will be proposed some individualized strategies. Types of intervention Depending on scores of motivation, the following strategies will be proposed to participants.

* identify the barriers related to physical activity
* increase informations related to physical activity and nutrition
* informations about the risk related to inactivity and diet
* ask to the individual to list and barriers related to barriers as thhe interest to modify the behavior.
* List persons who may act as social support
* set behavior change goals
* Increase self-confidence and self-efficacy about changing behavior
* Relaxation at home
* Use reinforcement management
* methods of time management
* counter-conditioning
* identify factors related to the relapse Time management Participants will be evaluated after the first 6 months. Then, they will be followed during 24 months. Statistical analysis Sample size The sample was calculated using a previous study. To obtain a difference of 0.51 in emotional eating with a standard deviation of 1.63 with an alpha risk of 5% and a power of 90%, the number of subject is 110 subject. Expected a drop-out of 20%, 138 subjects will be included. Predictive factors

  1. Identification of predictive factors Student T test to select the predictive factors
  2. Predictive factors Multiple linear regression
  3. Mechanisms analysis of mediation with the Baron and Kenny method

ELIGIBILITY:
Inclusion Criteria:

* Patients with obesity (grade 2 or 3)
* Age 18 to 65
* participation to the therapeutic training
* Patient with non physical activity

Exclusion Criteria:

* Patients needing chirurgigical act
* patient taking neuroleptic or psychiatric
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2013-11-22 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-11-12 (Actual)

PRIMARY OUTCOMES:
Emotional eating assessed by the Dutch Eating behavior questionnaire | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier-Hopital La colombière, Montpellier, France